CLINICAL TRIAL: NCT04472156
Title: A Prospective Study of a Mosaic Embryo Transfer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado Center for Reproductive Medicine (Other)
Responsible Party: Principal Investigator, Mandy Katz-Jaffe, Scientific and Genetics Director, Colorado Center for Reproductive Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mosaic
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Outcomes will be evaluated with women who have a mosaic embryo transferred
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transfer of mosaic embryo (Experimental): Women will have a mosaic embryo transferred to their uterus after in vitro fertilization (IVF) with pre implantation genetic testing completed at Colorado Center for Reproductive Medicine.
  Interventions: Procedure: Transfer of mosaic embryo

INTERVENTIONS:
Procedure: Transfer of mosaic embryo — Subjects will transfer a mosaic embryo transferred to their uterus

SUMMARY:
This research is a prospective study in which the purpose is to investigate the clinical outcomes following the transfer of a mosaic embryo (presence of both chromosomally normal and abnormal cells) that has been screened for preimplantation genetic testing (PGT).

DETAILED DESCRIPTION:
This research is a prospective study with the purpose is to investigate the clinical outcomes following the transfer of a mosaic embryo (presence of both chromosomally normal and abnormal cells) that has been screened for preimplantation genetic testing (PGT). PGT involves the biopsy and testing of a handful (3-6) of trophectoderm (pre-placental cells) from the embryo. Embryos that are screened as mosaic via PGT, as a standard, are not offered for transfer for pregnancy attempt. Publications have shown that mosaic embryos and mosaic fetuses can result in healthy live births (Wallerstein et al, 2015; Victor et al, 2019). Ongoing clinical outcomes are important to further understand the association between an embryonic mosaic biopsy of pre-placental cells and subsequent fetal chromosomal constitution. Implantation rates and live birth rates will be evaluated to help understand if mosaic embryos should routinely be offered for transfer to patients attempting pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Women age 18-45 Infertile women who have completed an IVF cycle with PGT at the Colorado Center for Reproductive Medicine (CCRM) that have a mosaic embryo
* Patients can be of any race, culture, sexual orientation or ethnicity
* Patients that are willing to transfer a single embryo

Exclusion Criteria:

* Patients that do not meet the clinical requirements for an embryo transfer per clinic standards.
* Patients that desire more than a single embryo transfer.
* Patients that are using a gestational carrier.
* Embryonic mosaic PGT results that include chromosome errors 13, 18, 21
* Patients that did not complete their IVF with PGT cycle at the Colorado Center for Reproductive Medicine.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 250 (Estimated)
Dates: Start 2020-10-15 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Implantation rate | 3-4 weeks after embryo transfer
  Ultrasound will be performed 2-3 weeks after initial positive pregnancy test to confirm viable pregnancy as evidenced by gestational sac in the uterus with a fetal heat rate
Live birth rate | 9-12 months post embryo transfer
  Live birth rate will be evaluated

SECONDARY OUTCOMES:
Miscarriage Rates | 5-12 months post embryo transfer
  The rate of miscarriage will be evaluated associated with a mosaic embryo transfer
Products of conception from miscarriage | 2-9 months post embryo transfer
  Products of conception will be karyotyped if available following a miscarriage and compared to that of previous PGT testing if the patient is willing to have the testing.
Pregnancy complications | 9-12 months post embryo transfer
  Patient will be evaluated after delivery to assess if patient had any complications associated with the pregnancy. This will be completed with telephone interview
Stillbirth rates associated with Mosaic Embryo Transfer | 9-12 months post embryo transfer
  The rate of stillbirths with will be evaluated among patients who have had a mosaic embryo transfer
Prenatal testing | 9-12 months post embryo transfer
  If available, we will request any results of prenatal testing of karyotype that was obtained via Amniocentesis or Chorionic Villa Sampling (CVS)
Neonatal Outcomes | 12-15 months after birth of baby
  Patient will be contacted to assess the health of the infant, noting any medical problems if any that the baby has.

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Katz-Jaffe, PhD, Principal Investigator — Fertility Genetics
Locations (1):
- Colorado Center for Reproductive Medicine, Lone Tree, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wallerstein R, Misra S, Dugar RB, Alem M, Mazzoni R, Garabedian MJ. Current knowledge of prenatal diagnosis of mosaic autosomal trisomy in amniocytes: karyotype/phenotype correlations. Prenat Diagn. 2015 Sep;35(9):841-7. doi: 10.1002/pd.4620. Epub 2015 Jun 23. PMID 25976239
- [Background] Victor AR, Tyndall JC, Brake AJ, Lepkowsky LT, Murphy AE, Griffin DK, McCoy RC, Barnes FL, Zouves CG, Viotti M. One hundred mosaic embryos transferred prospectively in a single clinic: exploring when and why they result in healthy pregnancies. Fertil Steril. 2019 Feb;111(2):280-293. doi: 10.1016/j.fertnstert.2018.10.019. PMID 30691630